CLINICAL TRIAL: NCT06868004
Title: Positive Impact of Holistic Nursing on Cognitive Impairment and Psychiatric Symptoms in Patients with Alzheimer's Disease
Brief Title: Holistic Nursing Benefits Cognitive and Psychiatric Symptoms in Alzheimer's Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First People's Hospital of Jingzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023199
Record Dates: First submitted 2025-03-05; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's Disease; Holistic nursing; Psychological state; Cognitive function; Psychiatric symptoms
MeSH Terms: conditions — Alzheimer Disease | interventions — Holistic Nursing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention)
- Observation Group (Experimental)
  Interventions: Behavioral: Holistic Nursing

INTERVENTIONS:
Behavioral: Holistic Nursing — The intervention in this study is based on Holistic Nursing (HN) for patients with Alzheimer's Disease (AD). It involves a comprehensive approach including psychological support, cognitive rehabilitation, memory enhancement, self-care training, and environmental modifications. Psychological interventions focus on personalized communication and emotional support, aiming to reduce negative emotions and improve trust in the healthcare team. Cognitive interventions include activities like painting, card recognition, and storytelling to enhance cognitive function. Memory interventions use personalized memory aids, and self-care interventions aim to improve daily living skills. The ward environment is adjusted to promote safety and comfort. This multi-faceted approach is designed to improve cognitive function, self-care abilities, and emotional well-being in AD patients.
  Arms: Observation Group

SUMMARY:
This clinical study aims to evaluate the effects of a holistic nursing (HN) intervention on cognitive function, psychological well-being, and overall health outcomes in patients with Alzheimer's disease (AD). AD is a progressive neurodegenerative disorder characterized by cognitive decline and behavioral changes, significantly impacting patients' quality of life and increasing the burden on caregivers. Conventional treatment primarily involves pharmacological interventions, but non-pharmacological approaches, such as specialized nursing care, have shown potential in improving patient outcomes.

This study prospectively enrolled 105 AD patients admitted to our hospital between January 2023 and January 2024. Patients were divided into two groups based on admission periods: the control group (n=58) received standard care, while the observation group (n=47) received HN in addition to standard care. The HN intervention was implemented based on established guidelines for older adults with cognitive impairment and consisted of five key components: psychological support, cognitive stimulation, memory enhancement, self-care training, and environmental optimization.

The study assessed cognitive function, psychiatric symptoms, anxiety, and depression levels before and after the intervention using validated scales, including the Mini-Mental State Examination (MMSE), Neuropsychiatric Inventory (NPI), Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-cog), Montreal Cognitive Assessment (MoCA), and Self-rating Anxiety/Depression Scales (SAS/SDS). Additionally, blood biomarkers related to neurological function, such as dopamine, acetylcholine, serotonin, γ-aminobutyric acid, S100β, homocysteine, and interleukin-1β, were measured.

Patient compliance, safety outcomes, and family satisfaction with the nursing intervention were also evaluated. The findings of this study may provide evidence supporting the integration of HN as a complementary approach in AD management, potentially improving cognitive function, reducing psychiatric symptoms, and enhancing overall patient well-being.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Alzheimer's Disease (AD) according to clinical and neuroimaging evidence.
* Aged between 60 to 80 years.
* Mild-to-moderate disease severity, with a Mini-Mental State Examination (MMSE) score ranging from 10 to 24.
* Adequate cognitive and functional capacity to complete questionnaires and follow the intervention protocol.
* Ability to communicate and comprehend instructions.
* Availability of comprehensive medical records.
* Informed consent obtained from the patient or their legal guardian.

Exclusion Criteria:

* History of intracranial surgery or major brain trauma.
* Coexisting psychiatric disorders or severe mental illnesses.
* Significant visual, auditory, language, or motor impairments that would hinder participation in the study.
* Severe organ dysfunction that could interfere with study participation or safety.
* Comorbid autoimmune diseases or severe malignancies.
* Participants who have received experimental treatments or clinical trials within the last 3 months.
* Pregnant or breastfeeding women.
* Individuals with a history of substance abuse or dependency.
* Participants with other medical conditions that, in the opinion of the investigator, would compromise participation in the study.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Change in Cognitive Function Assessed by MMSE | Baseline (before intervention) and after 6 months of intervention.
  The improvement in cognitive function will be measured using the Mini-Mental State Examination (MMSE) score. Cognitive changes will be evaluated pre- and post-intervention to assess the effectiveness of the Holistic Nursing intervention.
Change in Cognitive Function Assessed by MoCA | Baseline (before intervention) and after 6 months of intervention.
  The improvement in cognitive function will be measured using the Montreal Cognitive Assessment (MoCA) score. Cognitive changes will be evaluated pre- and post-intervention to assess the effectiveness of the Holistic Nursing intervention.

SECONDARY OUTCOMES:
Change in Psychiatric Symptoms Assessed by NPI | Baseline (before intervention) and after 6 months of intervention.
  Reduction in psychiatric symptoms will be measured using the Neuropsychiatric Inventory (NPI) score. Lower scores will indicate improvements in symptoms such as anxiety, depression, and agitation.
Change in Anxiety Levels (SAS Score) | Baseline (before intervention) and after 6 months of intervention.
  Anxiety levels will be measured using the Self-Rating Anxiety Scale (SAS). The SAS score ranges from 20 to 80, with higher scores indicating greater anxiety severity. A reduction in scores post-intervention will indicate an improvement in anxiety symptoms.
Medication Adherence | Baseline (before intervention) and after 6 months of intervention.
  Patient adherence to prescribed medication will be measured using the Morisky Medication Adherence Scale-8 (MMAS-8). The MMAS-8 score ranges from 0 to 8, with higher scores indicating better adherence to medication regimens.
Family Satisfaction | At discharge (approximately within 24 hours of patient discharge).
  Family satisfaction with nursing care and interventions will be assessed using a validated nursing satisfaction questionnaire. The questionnaire includes a Likert scale ranging from 1 to 5, where higher scores indicate greater satisfaction. The overall satisfaction rate will provide insights into the perceived effectiveness of the intervention from the family's perspective.
Change in Cognitive Function Related to Psychiatric Symptoms Assessed by ADAS-cog | Baseline (before intervention) and after 6 months of intervention.
  Cognitive changes associated with psychiatric symptoms will be measured using the Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-cog). Lower scores will indicate reduced cognitive impairment.
Change in Depression Levels (SDS Score) | Baseline (before intervention) and after 6 months of intervention.
  Depression levels will be measured using the Self-Rating Depression Scale (SDS). The SDS score ranges from 25 to 100, with higher scores indicating greater depression severity. A reduction in scores post-intervention will indicate an improvement in depression symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Jinzhou Medical University, Jinzhou, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yu J, Zhu L, Song Y, Shi B, Zhou X. Positive Impact of Holistic Nursing on Cognitive Impairment and Psychiatric Symptoms in Patients With Alzheimer's Disease. Actas Esp Psiquiatr. 2025 May;53(3):586-597. doi: 10.62641/aep.v53i3.1948. PMID 40355993